CLINICAL TRIAL: NCT02901002
Title: Body Perception and Complex Regional Pain Syndrome : a Case-control Study
Brief Title: Body Perception and Complex Regional Pain Syndrome
Acronym: SDRC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608097; 2016-A01248-43 (Other: ANSM)
Record Dates: First submitted 2016-09-05; First posted 2016-09-15 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2017-11

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Complex Regional Pain Syndromes; Pain; Spontaneous sensations; interoception
MeSH Terms: conditions — Complex Regional Pain Syndromes; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patients suffering from CRPS of the lower limb Patients with sensory testing in the two hand and neuropsychological evaluation
  Interventions: Other: Sensory testing in the two hand; Other: Neuropsychological evaluation
- Control: Healthy controls match by age, gender, Body Mass Index Healthy volunteers with sensory testing in the two hand and neuropsychological evaluation
  Interventions: Other: Sensory testing in the two hand; Other: Neuropsychological evaluation

INTERVENTIONS:
Other: Sensory testing in the two hand — spontaneous sensations while watching a hand
Other: Neuropsychological evaluation — Score to anxiety-depression scale

SUMMARY:
In CRPS, perturbation of body image and pseudo-neglect syndrome of the body part affected are frequently found. Pain and sensory perturbation seems to modify the way patients perceived their body part affected.

Does a local body image perturbation can affect the balanced of the global self-awareness?

DETAILED DESCRIPTION:
With the investigation of spontaneous sensations (SPS) according to the protocol of Michael and al (2011) the investigators study how patients can listen to their internal sensations located in other body part than the painful member in order to construct a representation of the body and maintain it in active consciousness. A group of controls will be included to understand if there is a global modification in the perception of SPS witch may be linked to the pathology.

ELIGIBILITY:
Inclusion Criteria:

* For patients:

  • a diagnosis of CRPS of the lower limb according to the Budapest Criteria (men or women) For patients and control group
* Age ≥ 18 years

Exclusion Criteria:

For patients and control group

* neurological disease with cerebral repercussion or not stabilized serious physical illness;
* psychotropic medication
* disorders related to the use of a psychoactive substance (abuse, dependence or withdrawal);

  * For patients:
* Presence of an other pain disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from CRPS of the lower limb and Healthy controls
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Sensory testing | day 1
  areas of the hand where spontaneous sensations were felt

SECONDARY OUTCOMES:
Neurological evaluation by questionary | day 1
  Score to HAD (anxiety-depression) scale

CONTACTS AND LOCATIONS:
Overall Officials: Christelle CREAC'H, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No